CLINICAL TRIAL: NCT00738478
Title: Phase III Study for the Significance of Nasogastric Decompression Tube After Curative Distal Gastrectomy for Gastric Cancer Patients
Brief Title: Quality of Life After Routine Nasogastric Decompression After Distal Gastrectomy for Gastric Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMC-RCTGastric01
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Cancer
Keywords: distal gastrectomy; quality of life
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Arm A: with nasogastric tube
  Interventions: Device: nasogastric tube
- B (Active Comparator): Arm B: without nasogastric tube
  Interventions: Device: without nasogastric tube

INTERVENTIONS:
Device: nasogastric tube — insertion of nasogastric tube for 2 days after operation
  Arms: A
Device: without nasogastric tube — without nasogastric tube after operation
  Arms: B

SUMMARY:
The aim of the study is to evaluate whether distal gastrectomy without post-operative nasogastric decompression tube is better in terms of quality of life.

DETAILED DESCRIPTION:
Nasogastric decompression tube is an intra-operative routine in most of the time to facilitate exposure of operative field during elective distal gastrectomy, however, whether it should be retained post-operatively is controversial. Nasogastric decompression tube helps to drain the gastric remnant in case there is edema around the gastrojejunostomy, ileus and delayed gastric emptying, which can theoretically relieve nausea and abdominal distension. However, nasogastric intubation could cause patients discomfort; also it has been shown that it would cause gastroesophageal reflux which may be associated with pulmonary complication.

ELIGIBILITY:
Inclusion Criteria:

* on the basis of whether distal gastrectomy was anticipated at WMUH for gastric cancer.

Exclusion Criteria:

* patients who were diagnosed inadequacy for this study by a physician.
* patients without an informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | seven days after operation

SECONDARY OUTCOMES:
complication, hematological data, | the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mikihito Nakamori, MD, Principal Investigator — Wakayama Medical University
Locations (1):
- Second Department of Surgery, Wakayama Medical University, Wakayama, Japan